CLINICAL TRIAL: NCT03243773
Title: Evaluation of Lung UltraSound In Acute Heart Failure (ELUSIA)
Brief Title: Evaluation of Lung Ultrasound in Acute Heart Failure
Acronym: ELUSIA
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Institutional Head, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Other Study IDs: BASEC 2015-00133
Record Dates: First submitted 2017-08-04; First posted 2017-08-09 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Acute Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard laboratory samples for blood cell count, blood chemistry including NT-proBNP
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Lung ultrasound — Point-of-care ultrasound exam of both lungs in 4 predefined zones.

SUMMARY:
Acute heart failure is a life threatening condition requiring rapid diagnosis and treatment. However, the differentiation between heart failure and other conditions presenting with acute dyspnea is notoriously difficult in the emergency room. Point-of-care lung ultrasound is a simple, rapid and noninvasive technique directly visualizing fluid content in the lung as evidence for acute heart failure. A number of publications showed the diagnostic utility of lung ultrasound in the diagnosis of heart failure, but many open questions remain.

The goal of this study is to evaluate the diagnostic accuracy of lung ultrasound to predict a cardiac origin of dyspnea in unselected patients in the emergency room as compared to standard evaluation. Further goals are to evaluate if lung ultrasound provides additional diagnostic information as compared to clinical examination, NT-proBNP and chest X-ray, to compare the diagnostic accuracy of lung ultrasound in different patient subgroups (heart failure with preserved vs reduced ejection fraction, de novo vs decompensated chronic heart failure, age ≥75 vs <75 years, women vs men and presence vs absence of concomitant pulmonary disease) and to compare demographics and clinical characteristics in different patient populations.

300 patients, aged ≥18 years presenting to the emergency room (ER) with acute dyspnoe as principal complaint will undergo initial clinical assessment of the likely etiology of dyspnea by the ER physician in charge. The second assessment by the same physician will include results of NT-proBNP according to predefined cutoffs. Final diagnosis ("Gold Standard") will be done by two experienced investigators after patient discharge taking into account the complete medical record except the results of lung ultrasound. Assessment of chest X-ray and lung ultrasound by investigators will be preforemd blinded regarding all other results.

DETAILED DESCRIPTION:
Evaluation of Lung Ultrasound in Acute Heart Failure (ELUSIA). A monocenter, randomised, double-blind, diagnostic clinical study.

Background and Rationale: Acute heart failure is a life threatening condition requiring rapid diagnosis and treatment. However, the differentiation between heart failure and other conditions presenting with acute dyspnea is notoriously difficult in the emergency room. Point-of-care lung ultrasound is a simple, rapid and noninvasive technique directly visualizing fluid content in the lung as evidence for acute heart failure. A number of publications showed the diagnostic utility of lung ultrasound in the diagnosis of heart failure, but many open questions remain.

Objective(s): 1) To evaluate the diagnostic accuracy of lung ultrasound to predict a cardiac origin of dyspnea in unselected patients in the emergency room as compared to standard evaluation. 2) To evaluate if lung ultrasound provides additional diagnostic information as compared to clinical examination, NT-proBNP and chest X-ray. 3) To compare the diagnostic accuracy of lung ultrasound in different patient subgroups (heart failure with preserved vs reduced ejection fraction, de novo vs decompensated chronic heart failure, age ≥75 vs <75 years, women vs men and presence vs absence of concomitant pulmonary disease. 4) To compare demographics and clinical characteristics in different patient populations.

Inclusion criteria: Emergency room presentation with acute dyspnoe as principal complaint (either new or worsening in the last 48 hours), age ≥18 years.

Exclusion criteria: Immediately life threatening condition (cardiac arrest, ST-elevation myocardial infarction, shock, respiratory failure requiring intubation), no consent.

Measurements and Procedures: Initial clinical assessment of the likely etiology of dyspnea by the emergency room physician in charge. Second assessment by the same physician including results of NT-proBNP according to predefined cutoffs. Final diagnosis ("Gold Standard") considering the complete medical record except the results of lung ultrasound by 2 experienced investigators after patient discharge. Assessment of chest X-ray and lung ultrasound by investigators blinded regarding all other results.

Study Product/Intervention: Point-of-care lung ultrasound in the emergency room as only study specific intervention. Registration of "B-lines" in 4 defined zones on both sides and calculation of a validated score. Digital storing of results for offline analysis.

Comparator(s): Comparison of the accuracy of lung ultrasound for the diagnosis of acute heart failure as compared to clinical investigation, NT-proBNP and chest X-ray alone or in combination.

Number of Participants: 300 patients. Based on the literature and clinical expericence we estimate than at least 50% of the patients will have a diagnosis of heart failure. In this group around 50% of patients will have heart failure with preserved, the other 50% with reduced ejection fraction. Most patients will suffer from decompensation of chronic heart failure and will be older than 75 years. Around 1/3 of the patients will have an additional diagnosis of chronic lung disease.

Study Duration: 3 years.

ELIGIBILITY:
Inclusion criteria:

Emergency room presentation with acute dyspnoe as principal complaint (either new or worsening in the last 48 hours) Age ≥18 years.

Exclusion criteria:

Immediately life threatening condition (cardiac arrest, ST-elevation myocardial infarction, shock, respiratory failure requiring intubation) No consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected patients presenting with this acute dyspnea to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Value of lung ultrasound in the diagnosis of acute heart failure | at the time of inclusion into the study
  Presence/Absence of heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rickenbacher, MD, Principal Investigator — Cantonal Hospital Baselland
Locations (1):
- Cantonal Hospital Baselland, Bruderholz, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No